CLINICAL TRIAL: NCT03798028
Title: The Effects and Safety of Mesenchymal Stem Cells in the Treatment of Moderate/Severe Rheumatoid Arthritis， a Multicenter Randomized Controlled Clinical Study
Brief Title: The Safety and Effects of Mesenchymal Stem Cell (MSCs) in the Treatment of Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: Changhai Hospital (Other); Southwest Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014ZX09508002
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2018-12

CONDITIONS: Rheumatoid Arthritis
Keywords: anemia; Interstitial pulmonary disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Anemia; Lung Diseases, Interstitial

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UC-MSCs treatment (Experimental): the participants will receive the single-dose UC-MSCs (1×10^6 cells/kg ) in combined with the present treatment.
  Interventions: Biological: UC-MSCs
- no UC-MSCs treatment (No Intervention): the participants will receive the placebo in combined with the present treatment.

INTERVENTIONS:
Biological: UC-MSCs — The UC-MSCs will be administrated by intravenous injection at the dose of 1×10^6 cells/kg.
  Other Names: placebo
  Arms: UC-MSCs treatment

SUMMARY:
This study evaluates the safety and therapeutic effects of single-dose human umbilical cord blood mesenchymal stem cells (UC-MSCs) on the adult patients with moderate/severe Rheumatoid Arthritis accompany with anemia or/and Interstitial pulmonary disease. Half of participants will receive UC-MSCs and keep the present medication,while the other half will receive a placebo and keep the present medication.

ELIGIBILITY:
Inclusion Criteria:

1. Fulfill 2010 ACR/ the European League Against Rheumatism (EULAR) classification criteria or the 1987 ACR classification criteria.
2. Age limits:18 to 70 years old.
3. Freely given informed consent.
4. Disease Activity Score (DAS) 28≥3.2或 Simple Disease Activity Index (SDAI)>11.0或 Clinical Disease Activity Index (CDAI) >10.0.
5. Hemoglobin < 90 g/L and/or interstitial lung disease shown in high resolution CT.
6. Poor response to current treatment. The current treatment refers to receive the medicines (including Leflunomide, Methotrexate, Sulphasalazine, Hydroxychloroquine, Cyclosporine A,and Tacrolimus, alone or in combination ) for 3 months, and maintain the stable-dose of drugs for at least 1 month.
7. More than 3 months and a stable dose for at least 1 month are required if glucocorticoid is used. The dose of glucocorticoid is less than or equal to10mg/ day of prednisone.

Exclusion Criteria:

1. Participants who received glucocorticoid therapy by intra-articular injection within 1 week.
2. Glucocorticoid that participants received is more than 10 mg/day of prednisone within 1 months.
3. Complication with other connective tissue disease (except for Sjogren syndrome) .
4. Participants with chronic and acute infection (bacteria, virus and parasite,etc.).
5. Participants with acute and chronic tuberculosis infection.
6. Malignant tumors or participants with a family history of malignant tumors.
7. Participants have a family history of allergic conditions.
8. Participants infected by Hepatitis B Virus(HBV), Hepatitis C Virus (HCV) and Human Immunodeficiency Virus （HIV）.
9. Participants suffer from central nervous system demyelinating disease or multiple sclerosis (MS) currently or in the past.
10. Participants received live vaccines with 3 months.
11. Drug abuse and alcoholism.
12. Participants with severe mental or neurological disorders that affect informed consent and/or the presentation or observer of adverse events.
13. Participants with pregnant or in breast-feeding, and patients who has a pregnancy plan within 1 year.
14. Participants received stem cell therapy in the past.
15. Participants received any biological agents within 3 months.
16. Anemia (such as anemia with dysplasia) and interstitial lung disease for other reasons.
17. Participants with cardiovascular and cerebrovascular damage, such as thrombosis.
18. Participants taking drugs that affect the test for blood and lung.
19. Participants taking any traditional Chinese medicine.
20. Participants taking immune modulators such as Transfer Factor, Thymosin and Intravenous Immunoglobulin (IVIG), and so on.
21. Other cases that participants are considered by investigator that they did not meet the requirements for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2017-12-26 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Improvement rate of blood routine hemoglobin (HGB) compared to baseline. | 24 weeks
  The HGB increases by 10g compared to the baseline is considered improvement.
Improvement rate of forced vital capacity (FVC) and/or carbon monoxide diffusing capacity (DLCO) compared to baseline. | 24 weeks
  FVC increases by 0.5% and DLCO increases by 10% compared to baseline are considered improvement.

SECONDARY OUTCOMES:
The remission rates of American College of Rheumatology (ACR) 20, ACR 50 and ACR 70. | 12 weeks and 24 weeks
  The patients achieves 20%, 50%, or 70% remission according to American College of Rheumatology (ACR) criteria.
White blood cell count and platelet count improved compared to the baseline. | 12 weeks and 24 weeks
  White blood cell count increases to the 3.5×10^9/L and platelet count increases to 80×10^ 9.
Improvement rate of blood routine hemoglobin (HGB) compared to baseline. | 12 weeks
  The HGB increases by 10 g compared to the baseline is considered improvement.
Improvement rate of forced vital capacity (FVC) and/or carbon monoxide | 12 weeks
  FVC increases by 0.5% and DLCO increases by 10% compared to baseline
Image improvement of lung on high resolution CT. | 24 weeks
  The area change of image of lung.
Improvement of 6-minute walking distance compared to baseline. | 12 weeks and 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China